CLINICAL TRIAL: NCT00576173
Title: An Open Label Study to Evaluate Safety, Tolerability and Clinical Utility of ULTRACET® (37.5mg Tramadol Hydrochloride/325mg Acetaminophen) for the Treatment of Breakthrough Pain in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014683
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: Cancer pain; Breakthrough pain; acetaminophen; tramadol hydrochloride; Ultracet
MeSH Terms: conditions — Pain; Cancer Pain; Breakthrough Pain | interventions — Ultracet

INTERVENTIONS:
Drug: tramadol hydrochloride; acetaminophen

SUMMARY:
The purpose of this study is to evaluate the analgesic effectiveness and safety of 37.5mg Tramadol hydrochloride/325mg Acetaminophen in the treatment of breakthrough pain in cancer patients.

DETAILED DESCRIPTION:
The combination of tramadol HCI/acetaminophen provides a more rapid onset of action compared to tramadol HCI alone and a longer duration of action than acetaminophen alone. Therefore, the combination of tramadol and acetaminophen may be effective for the treatment of cancer pain as well as to allow lower cumulative daily dosages of each medication to be used.This is an open-label study. Patients will receive one-dose treatment of 37.5mg Tramadol/325mg Acetaminophen tablets.This study has been designed to investigate the following hypothesis:Tramadol hydrochloride/acetaminophen is effective in the treatment of breakthrough pain in cancer patients.The patients will complete basic questions on side effect at visits on entry, 10, 30 mins, and 1h.

The patients will receive only one dose treatment of Tramadol hydrochloride/Acetaminophen oral tablets throughout the study. The number of oral tablets be given will be depend on the total daily dose of around-clock medications. If around-clock medication is Tramadol <=400mg or codeine <=300mg or morphine <60mg, the breakthrough pain medication will be 1 tablet. If around-clock medication is morphine 60-120mg or Fentanyl >=25 ug/hr, the breakthrough pain medication will be 2 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically, radiologically or haematologically confirmed malignancy whose pain is judged by the investigator to be caused by the malignancy
* Patients must have been on a stable daily dose of weak opioids or strong opioids for at least 72 hours prior to the start the study and must remain at the same dosage for the duration of the study
* Patients must have a VAS (Visual analog scale) >=40mm

Exclusion Criteria:

* Patients who have taken either morphine with daily dose more than 120mg or Fentanyl with daily dose more than 50ug/hr
* Patients with significant abnormalities in hepatic or renal function which would, in the opinion of the investigator, prevent the patients involvement in the study
* Patients with significant clinical abnormalities in CNS, respiratory or cardiovascular function, which in the investigators judgement prevents participation in the study
* Patients who have taken antidepressants or anti-epileptic drugs, sedative hypnotics, selective serotonin reuptake inhibitor, short-acting analgesics, topical medications and anesthetics and/or muscle relaxants when taking Tramadol/Acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity and side effect will be assessed on entry, 10, 30 mins, and 1hour. In addition, the amount of rescue analgesic medication consumed will be recorded by the patient and summarized by the investigator at study visits.

SECONDARY OUTCOMES:
Investigator global assessment and patient global assessment for the treatment with respect to pain control, side effects and overall using a 5-point scale at the end of the treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd